CLINICAL TRIAL: NCT03036644
Title: Effects of Electronic Cigarette Vaporization at High Temperature in Comparison to Tobacco Smoking on Cardiovascular Function and Oxidative Stress in Electronic Cigarette Users and Regular Tobacco Smokers
Brief Title: Comparison of Electronic Cigarettes and Tobacco Cigarettes on Cardiovascular Function and Oxidative Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Martin Chaumont, Principal investigator, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: P2017/028 / B406201630672
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Risk Factor
Keywords: electronic cigarette; e-cigarette; oxidative stress; tobacco smoking
MeSH Terms: conditions — Vaping; Tobacco Smoking | interventions — Tobacco Use Cessation Devices; Diathermy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- e-cigarette nic_O LT (Experimental): e-cigarette (without nicotine; low temperature)
  Interventions: Device: e-cigarette (PG+VG without nicotine; low temperature)
- e-cigarette Nic_1 LT (Experimental): e-cigarette (with nicotine; low temperature)
  Interventions: Device: e-cigarette (PG+VG with nicotine; low temperature)
- e-cigarette Nic_0 HT (Experimental): e-cigarette (without nicotine; high temperature)
  Interventions: Device: e-cigarette (PG+VG without nicotine; high temperature)
- e-cigarette NIC_1 HT (Experimental): e-cigarette (with nicotine; high temperature)
  Interventions: Device: e-cigarette (PG+VG with nicotine; high temperature)
- Tobacco cigarette (Active Comparator): Tobacco cigarette
  Interventions: Other: tobacco cigarette
- Placebo (Placebo Comparator): No E-cigarettes, Nor tobocco cigarettes
  Interventions: Device: e-cigarette (PG+VG without nicotine; low temperature)

INTERVENTIONS:
Device: e-cigarette (PG+VG without nicotine; low temperature)
  Arms: Placebo; e-cigarette nic_O LT
Device: e-cigarette (PG+VG with nicotine; low temperature)
  Arms: e-cigarette Nic_1 LT
Device: e-cigarette (PG+VG without nicotine; high temperature)
  Arms: e-cigarette Nic_0 HT
Device: e-cigarette (PG+VG with nicotine; high temperature)
  Arms: e-cigarette NIC_1 HT
Other: tobacco cigarette
  Arms: Tobacco cigarette

SUMMARY:
Background: Electronic cigarettes (e-cigarettes) are battery-powered devices heating a liquid (e-liquid) composed of propylene glycol and/or vegetable glycerin, and most commonly, nicotine to form an aerosol (vapor) that is inhaled (i.e. "vaped"). Scarce and conflicting data are available regarding the cardiovascular toxicity of e-cigarettes. We wish to determine the acute effects of propylene glycol/vegetable glycerin and nicotine vaporization at high temperature in comparison to tobacco cigarette smoking on several advanced cardiovascular parameters in healthy chronic e-cigarettes users and tobacco smokers. Furthermore, a large range of plasma, urine and respiratory oxidative stress markers will be quantified. By this way, we aim to demonstrate that e-cigarettes-induced systemic oxidative stress could be linked to cardiovascular toxicity. To the best of our knowledge, this is the first project that evaluates the effects of e-cigarettes vaping in comparison to tobacco cigarette smoking on the cardiovascular system in relation to vaporization temperature, nicotine delivery and oxidative stress.

Aims of the study: This study tests the following hypotheses: 1) acute high temperature vaporization of propylene glycol and vegetable glycerin has no deleterious effects on cardiovascular parameters in comparison to tobacco smoking; 2) Tobacco smoking rises plasma and urine oxidative stress biomarkers. On the contrary, acute and chronic e-cigarettes vaping don't rise these biomarkers. At a cellular level, plasma of smokers but not vapers increases superoxide anion production.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of pulmonary disease like asthma or COPD
* Any form of systemic or chronic disorder
* Active allergy within 4 weeks of the study
* Symptoms of infection or inflammation within 4 weeks of the study
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in subcutaneous flux | 1 hour

SECONDARY OUTCOMES:
Change in Plasma and urine oxidative stress markers | 1 hour
Change in aortic stiffness | 10 minutes
Change in heart rate variability | 10 minutes
Change in baroreflex sensitivity | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul Van Vooren, Study Director — Hospital Erasme
Locations (1):
- Erasme Hospital, Brussels, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chaumont M, Bernard A, Pochet S, Melot C, El Khattabi C, Reye F, Boudjeltia KZ, Van Antwerpen P, Delporte C, van de Borne P. High-Wattage E-Cigarettes Induce Tissue Hypoxia and Lower Airway Injury: A Randomized Clinical Trial. Am J Respir Crit Care Med. 2018 Jul 1;198(1):123-126. doi: 10.1164/rccm.201711-2198LE. No abstract available. PMID 29451806